CLINICAL TRIAL: NCT00569608
Title: Early Discharge Program From a Regional Reference Neonatal Intensive Care Unit
Brief Title: Early Hospital Discharge Program in Neonatology
Acronym: EDNEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Para La Investigacion Hospital La Fe (Other)
Responsible Party: JOSE LUIS CASTELL RIPOLL, FUNDACION INVESTIGACION HOSPITAL LA FE
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: FIHLaFe; AP015/06
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2005-06

CONDITIONS: Prematurity
Keywords: Parental stress; Early discharge; Anxiety; Depression; Neonatal Intensive Care Unit
MeSH Terms: conditions — Premature Birth; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EDA (Experimental): Neonates submitted to the protocol of early discharge.
  Interventions: Other: Early Discharge
- SDP (No Intervention): Discharge following the standard protocol of the neonatal intensive care unit.

INTERVENTIONS:
Other: Early Discharge — Application of an early discharge protocol from the neonatal intensive care unit.
  Arms: EDA

SUMMARY:
Early discharge of premature infants from the Neonatal Intensive Care Unit will have substantial benefits:

(i) diminish parental stress;

(ii) increase parental - child bonding;

(iii) diminish medical complications derived from prolonged hospitalization;

(iv) reduce cost;

(v) increase number of point of attendance disponible for future patients.

DETAILED DESCRIPTION:
Extremely premature infants have to remain for very prolonged time in the hospital. As a consequence, difficulties for establishing an adequate parental-infant bonding arise causing a substantial parental stress manifested as anxiety and depression, and increasing the risk of short and longterm consequences (neglect, abuse, maltreatment, abandonment). In addition, prolonged hospital stay will increase the probability of having medical complications (infections, excessive blood tests or image studies) and the cost of staying. Once the baby has improved sufficiently early discharge may be given independently of the baby's weight. In order to be successful, caregivers, psychologist and parents have to put forward an established protocol to be able to face satisfactorily this situation. We hypothesize that, with an adequate Early Discharge Program, we could substantially reduce length of hospitalization, cost, and reduce parental stress.

ELIGIBILITY:
Inclusion Criteria:

* Prematurity
* No need for hospital support
* Parents fulfill sociological score
* Cooperation of primary care pediatrician

Exclusion Criteria:

* Active disease
* Need for hospital intervention
* Major congenital malformations
* Chromosomopathies

Ages: 36 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2005-01; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Reduction in the length of hospitalization. | Days of hospitalization

SECONDARY OUTCOMES:
Parental stress | up to 3 months post discharge
Use of Health Resources of the Community | up to 3 months post discharge
Reduction in cost of hospitalization | Reduction in euros/baby

CONTACTS AND LOCATIONS:
Overall Officials: PILAR SAENZ, MD, Study Director — AGENCIA VALENCIANA DE SALUT
Locations (1):
- Hospital Universitario La Fe, Valencia, Spain

REFERENCES:
- [Result] Psychological distress in parents of premature infants at discharge from the nicu. Saénz P1, Cerdá M1, Gorba M1, Díaz Cordobés JL2, Yi, P2, Barreto, P2 ;Vento M (Sponsored by Maximo V, Prof)1Servicio de Neonatología, Hospital Universitario Materno Infantil La Fe, Valencia, Spain and 2Departamento de Personalidad, Evaluación y Tratamientos Psicológicos., Facultad de Psicología., Valencia, Spain. EPAS 2007; 616280.26
- [Result] Psychological follow up of parents of preterm infants enrolled in an early discharge program from the nicu. Saénz P1, Díaz Cordobés JL2, Cerdá M1, Boronat N1, Barreto P2, Yi P2; Vento M1. (Sponsored by Maximo Vento,)1Servicio de Neonatología, Hospital Universitario Materno Infantil La Fe, Valencia, Valencia, Spain and 2Dpto Personalidad, Evaluación y Tratamientos Psicológicos, Faculty of Psychology (University of Valencia), Valencia, Valencia, Spain. EPAS 2007; 616280.27
- [Result] Vulnerability Of Parents Of Very Low Birth Weight Infants (Vlbw) During Nicu Hospitalization. Saénz P1, Díaz Cordobés JL2, Cerdá M1, Boronat N1, Yi P2, Barreto P2 ; Vento M1. (Sponsored by Maximo Vento, Prof)1 Servicio de Neonatología, Hospital Universitario Materno Infantil La Fe, Valencia, Valencia, Spain and 2Departamento de Personalidad, Evaluación y Tratamientos Psicológicos., Facultad de Psicología.Universidad de Valencia., Valencia, Valencia, Spain. EPAS 2007; 618442.13
- [Derived] Saenz P, Cerda M, Diaz JL, Yi P, Gorba M, Boronat N, Barreto P, Vento M. Psychological stress of parents of preterm infants enrolled in an early discharge programme from the neonatal intensive care unit: a prospective randomised trial. Arch Dis Child Fetal Neonatal Ed. 2009 Mar;94(2):F98-F104. doi: 10.1136/adc.2007.135921. Epub 2008 Jul 17. PMID 18635681